CLINICAL TRIAL: NCT05210296
Title: The Effect of Lower Extremity Strengthening Exercises Versus Trunk Strengthening Exercises on Balance and Gait Functions in Elderly Individuals
Brief Title: The Effect of Lower Extremity Strengthening Exercises Versus Trunk Strengthening Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Fahri Köroğlu, Lecturer, Physiotherapist, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YALOVAÜNİVERSİTESİ-FAHRİ.K-077
Record Dates: First submitted 2021-12-25; First posted 2022-01-27 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Elderly; Balance; Gait
Keywords: Elderly; Gait Functions; Balance; Strengthening Exercises; Trunk
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trunk strengthening exercises (Experimental): After 5 minutes of warm-up exercises, 20 minutes of trunk strengthening exercises and 10 minutes of balance exercises will be applied to the participants, and the session will end with 5 minutes of cooling-off exercises.
  In trunk strengthening exercises, trunk resistance exercises will be applied with an elastic exercise band.
  Interventions: Behavioral: Exercises
- Lower extremity strengthening exercises (Experimental): After 5 minutes of warm-up exercises, lower extremity strengthening exercises and 10 minutes of balance exercises will be applied to the participants, and the session will end with 5 minutes of cool-down exercises.
  In lower extremity strengthening exercises, lower extremity resistance exercises will be applied with elastic exercise band.
  Interventions: Behavioral: Exercises
- Control (No Intervention): Participants will not be included in any exercise program. At the end of the study, the elderly will be informed about the effects of exercises and appropriate exercise program training will be given.

INTERVENTIONS:
Behavioral: Exercises — Therapeutic exercise will be applied to the elderly
  Arms: Lower extremity strengthening exercises; Trunk strengthening exercises

SUMMARY:
The aim of this study is to investigate the effect of lower extremity strengthening exercises versus trunk strengthening exercises on balance, walking, fall risk and quality of life in elderly individuals. In our study, the participants will be divided into 3 groups consisting of trunk strengthening exercises, lower extremity strengthening exercises and control groups.Body strengthening exercises and lower extremity strengthening exercises group will be included in the exercise program for a total of 40 minutes each session, 3 sessions a week, for a total of 8 weeks. The exercises will be shown and applied by the research physiotherapist in groups of 2-3 to the participants of both groups. No exercise program will be applied to the control group, and appropriate exercise training will be given after the final evaluation.

DETAILED DESCRIPTION:
Those aged 65 and over, residing in Yalova and agreeing to be included in the study, will be included in the study. Volunteers who will participate in the study will be informed about the purpose of the study, its duration, and possible side effects of the treatment to be applied. Their consent will be obtained with an "Informed Consent Form" prepared in accordance with the standards determined by the Clinical Research Ethics Committee of Istanbul University Cerrahpaşa Faculty of Medicine, and the study will be carried out in accordance with the Declaration of Helsinki. In our study, the participants will be divided into 3 groups consisting of trunk strengthening exercises, lower extremity strengthening exercises and control groups.

Body strengthening exercises and lower extremity strengthening exercises group will be included in the exercise program for a total of 40 minutes each session, 3 sessions a week, for a total of 8 weeks. The exercises will be shown and applied by the research physiotherapist in groups of 2-3 to the participants of both groups. No exercise program will be applied to the control group, and appropriate exercise training will be given after the final evaluation.

Evaluation scales will be administered to the participants at the beginning of the study and 8 weeks later.

Body weight, own weight of the extremity and elastic exercise band will be used in strengthening exercises in trunk strengthening exercises and lower extremity strengthening exercises groups.

The weight of the extremity itself, or the number of repetitions in exercises using body weight, will be determined at the initial assessment according to the patient's exercise tolerance for each exercise. For each exercise, the exercise program will be started with the number of repetitions perceived by the participant according to the Modified Borg Scale (MBS), the number of repetitions will be increased, the program will be continued with the number of repetitions, the perceived fatigue severity will be between 4-7, by increasing the number of repetitions weekly. will be.

Appropriate band selection for the exercises to be used with an elastic exercise band will be determined according to the participant's tolerance and muscle strength. Participants will be asked to do the exercise for 15 repetitions with the lowest level of exercise band first, and then the perceived fatigue severity will be questioned by MBS. If the exercise intensity perceived by the participant is between 4 and 7, it will be determined as the correct band. If the participant's perceived severity is lower, the process with the next higher band will be repeated until the correct band is found for the patient. The same process will be applied for the tape to be used in the strengthening training of each region.

Elastic band exercises will be started with 8 repetitions, and the intensity of exercise will be questioned by increasing the number of repetitions by 2 in the first exercise session each week. If the perception of exercise intensity has increased, the number of repetitions will be kept the same, if the exercise intensity does not increase, the number of repetitions will be continued as 10, the next week after the exercise as 12 repetitions, the color of the exercise band will be changed and the exercise intensity will be evaluated by switching to the next band, and if the exercise intensity is appropriate, the previous band will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Having adequate cognitive function ((Mini Mental State Test (MMST) score equal to or greater than 24)
* Functional Ambulation Classification (FAC) level of 3, 4 or 5.

Exclusion Criteria:

* Having cardiac diseases that prevent exercise
* Have had any cardiac event or surgery in the last six months
* Pulmonary embolism and deep vein thrombosis in the last three months
* History of disabling cerebrovascular disease
* Presence of acute retinal hemorrhage or previous ophthalmic surgery
* Presence of active infection, malignancy or multiple organ failure
* Terminal disease status
* Having a history of lower and upper extremity fractures in the last three months
* Severe hearing and vision loss
* Being diagnosed with Parkinson's, dementia, or depression
* Have received exercise training in the last six months
* Multiple drug use
* Having been diagnosed with vestibular disease
* Existence of moderate or severe respiratory system disease that is not under control that interferes with exercise
* Having uncontrolled hypertension
* Having diabetes with diabetes complications such as nephropathy, retinopathy and severe neuropathy, or uncontrolled diabetes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Balance Evaluation Systems Test (Mini BESTest) | 8 weeks
  It is a test developed by using factor analysis to determine the most important elements that represent dynamic balance, and the insensitive elements other than these are eliminated. It is a reliable assessment method that provides information on which balance systems are impaired in older adults. It includes tasks in the subsections "Forward-looking", "Reactive postural control", "Sensory orientation" and "Dynamic walking" and consists of 14 items scored from 2 (normal) to 0 (severely deficient). A total of 28 points can be obtained, higher scores indicate better balance
Activity-Specific Balance Confidence Scale | 8 weeks
  The scale includes 16 parameters related to exterior and interior spaces in daily living activities. It assesses the perception of balance and fear of falling. Balance confidence is scored between 0-100%. It is an easy-to-apply scale that can be completed in as little as 5 minutes.
Dynamic Gait Index | 8 weeks
  It is a test that measures the capacity to adapt to changes during walking. It evaluates activities such as slow walking, fast walking, walking with head movements, turning, climbing stairs, jumping obstacles, 0 points weak and 3 points successful. Low scores that can be obtained from the scale are indicative of disorders that may cause falls. Evaluates a total of 8 parameters over 24 points. A score of nineteen and below defines the presence of fall risk.

SECONDARY OUTCOMES:
Trunk Muscle Strength Measurement | 8 weeks
  For the measurement, they are asked to push the handheld dynamometer held steady for five seconds with all their strength. Trunk flexor, extensor, right and left lateral flexor, right and left rotator muscle strength will be evaluated. The measurement score will be taken as the highest value test score out of three measurements made two minutes apart.
Lower Extremity Muscle Strength Measurement | 8 weeks
  For the measurement, they are asked to push the handheld dynamometer held steady for five seconds with all their strength. Muscle strength of lower extremity hip flexor-extensor-abductors, knee flexors and extensors, ankle dorsi and plantar flexors will be evaluated. The measurement score will be taken as the highest value test score out of three measurements made two minutes apart.
10 Meter Walk Test | 8 weeks
  In this test, the person is asked to walk at their own normal pace in a pre-measured 10 meter area (if using walking aid, it will be carried out with it). The time starts when the person's foot is on the starting line and ends when he crosses the finish line. Two measurements are made and the best value is recorded in meters/second (m/s).
Tinetti Balance and Gait Test (TBGT) | 8 weeks
  TBGT, which is preferred especially in determining the risk of falling in the elderly, was first developed by Mary Tinetti under the name Performance-Oriented Assessment of Mobility Problems in Elderly Patients to evaluate patients at high risk of falling. It was later developed and named Tinetti Gait and Balance Assessment. TBGT evaluates balance ability and gait under 2 main headings: The first 9 items are about balance and the next 7 items are about walking. The total score of the first 9 items gives the balance score, and the total score of the next 7 items gives the walking score. If the total score of the scale is 18 and below, the risk of falling is high, if it is 19-24, the risk of falling is moderate, and a score of 25 and above indicates a low risk of falling.
Nottingham Health Profile (NHP) | 8 weeks
  NHP is a measure of general health status that measures individuals' perceived distress in physical, emotional and social areas. It consists of a total of 38 items: physical mobility (8 items), pain (8 items), sleep (5 items), emotional reactions (9 items), social isolation (5 items) and energy level (3 items). Each item is answered as "yes" or "no". It is one of the advantages of the scale that it includes sleep and pain sub-headings, and it allows a versatile assessment of the individual's point of view on health.

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)